CLINICAL TRIAL: NCT02789540
Title: An Observational, Multinational, Cross Sectional Primary Data Collection Study to Describe Symptoms Around 24-hs and Their Relationship With Adherence to Respiratory Treatment, Direct Costs and Patient Reported Outcomes (PRO) in Stable COPD Patients in Latin America.
Brief Title: Latin American Study of 24-hs Symptoms in Chronic Obstructive Pulmonary Disease (COPD) Patients; LASSYC Study
Acronym: LASSYC
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00112
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Stable COPD Patients
Keywords: COPD symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-country, multicentre, observational prospective data collection cross sectional study of patients with stable COPD in Latin America. Primary objective is to assess and characterize COPD symptoms over a period of 24 hours, by collecting information about the respiratory symptoms experienced at different times of the day and night-time in patients with stable COPD under real clinical practice conditions. Correlation between each of these symptoms and the Global Initiative for Chronic Obstructive Lung Disease (GOLD) classification, adherence to respiratory treatment, level of dyspnea, disease severity, comorbidities and physical activity as well direct costs will be done as secondary objectives. Study population are patients of 40 years and older, smokers or ex smokers of >= 10 pack/years with previous COPD diagnosis, attending outpatient specialists consults in Argentina, Chile, Colombia, Uruguay, Costa Rica, Guatemala and Mexico. Sample size is targeted to 900 enroled patients in order to ensure 860 patients to achieve statistical power to primary objective.

DETAILED DESCRIPTION:
This is a multi-country, multicentre, observational prospective data collection cross sectional study of patients with stable COPD in Latin America. Primary objective is to describe prevalence, severity and interrelationship of early morning, day and night-time symptoms in patients with stable COPD in Latin America (LatAm). Secondary objectives are to evaluate the relationship between early morning, day and night-time symptoms and 2013 GOLD classification, adherence to respiratory treatment (TAI and Morisky Medicaction Adherence Scale - MMAS-8), level of dyspnea (mMRC), disease severity (BODEX), comorbidities (COTE) and physical activity (IPAQ) as well direct costs by assessing health resources utilization (HRU) and exacerbations during last 12 months and respiratory treatment of last 2 months. Study population are patients of 40 years and older, smokers or ex smokers of >= 10 pack/years with previous COPD diagnosis, attending outpatient specialists consults in Argentina, Chile, Colombia, Uruguay, Costa Rica, Guatemala and Mexico. Sample size is targeted to 900 enroled patients in order to ensure 860 patients to achieve statistical power to primary objective. Data source and study conduct: site staff will retrospectively collect the necessary information from the patient's medical record to determine eligibility. Consecutively, patients with diagnosis and stable COPD will be screened and, if eligible, consented and enrolled. There will be only one study visit. For each patient, the physician will collect the following data at visit (from medical records or interviewing in study visit): social demographics, health insurance system, lifestyle, smoking history, comorbidities, level of dyspnea, disease severity, COPD prescribed treatments including therapeutic class, device, modality (rescue/maintenance) and posology during last past 2 months, exacerbations history and healthcare resources utilisation during last 12 months. In addition, the patient will be asked to provide data on disease-related symptomatology assessed during 24 hs day (early morning, daytime and night time symptoms), adherence to inhalers, health-related quality of life (HRQoL) and physical activity. AstraZeneca will develop Data Management Plan (DMP) and a website database platform for the purpose of this study. Data will be registered by PI directly in a website data platform. The LASSYC study is an observational cross sectional study which does not involve or study a specific medicinal product. Because of the non-interventional nature of this study, a simple monitoring plan is required. 100% of source data verification (SDV) of 10% of total enrolled patients, estimating that one site per country would be enough.The Non-Interventional Study will be performed in accordance with ethical principles that are consistent with the Declaration of Helsinki, International Conference on Harmonization (ICH)and Good Clinical Practice (GCP) and the applicable legislation on Non-Interventional Studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 40 years or older.
* Patient has diagnosis of COPD for 1 year or more.
* Patient has at least one spirometry with COPD criteria, fixed ratio <0.70 post bronchodilators (BD), in previous 12 months
* Patient is a current smoker or an ex-smoker with a smoking history of ≥ 10 pack-years.
* Stable patients, as stated in medical records or patient reports during visit, defined as: without exacerbation treatment at study visit neither in the previous 2 months, and without changes in maintenance COPD treatment regimen over the preceding 2 months (avoid first consult patient)
* Patients must be able and willing to read and comprehend written instructions, and comprehend and complete the questionnaires required by the protocol
* After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.

Exclusion Criteria

* Patient has diagnosis of sleep apnea syndrome or other chronic respiratory disease different from chronic obstructive diseases.
* An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to complete questionnaires or participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of 40 years and older, smokers or ex smokers of >= 10 pack/years with previous COPD diagnosis, attending outpatient specialists consults in Argentina, Chile, Colombia, Uruguay, Costa Rica, Guatemala and Mexico
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-06-10 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of daily COPD symptoms | Day one
  E-RS Questionnaire
Prevalence and severity of early morning COPD symptoms | Day one
  EMSCI Questionnaire
Prevalence and severity of night-time COPD symptoms | Day one
  NiSCI Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marc Miravitlles, MD, PhD, Study Chair — Hospital Universitari Vall d'Hebron. Barcelona
Locations (6):
- Research Site, Buenos Aires, Argentina
- Research Site, Santiago, Chile
- Research Site, Bogotá, Colombia
- Research Site, San José, Costa Rica
- Research Site, Mexico City, Mexico
- Research Site, Montevideo, Uruguay

REFERENCES:
- [Derived] Miravitlles M, Menezes A, Lopez Varela MV, Casas A, Ugalde L, Ramirez-Venegas A, Mendoza L, Lopez A, Wehrmeister FC, Surmont F, Montes de Oca M. Prevalence and impact of respiratory symptoms in a population of patients with COPD in Latin America: The LASSYC observational study. Respir Med. 2018 Jan;134:62-69. doi: 10.1016/j.rmed.2017.11.018. Epub 2017 Nov 28. PMID 29413510
- [Derived] Montes de Oca M, Menezes A, Wehrmeister FC, Lopez Varela MV, Casas A, Ugalde L, Ramirez-Venegas A, Mendoza L, Lopez A, Surmont F, Miravitlles M. Adherence to inhaled therapies of COPD patients from seven Latin American countries: The LASSYC study. PLoS One. 2017 Nov 15;12(11):e0186777. doi: 10.1371/journal.pone.0186777. eCollection 2017. PMID 29140978
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4132&filename=Resumen_Resultados_LASSYC.pdf